CLINICAL TRIAL: NCT03514966
Title: Repetitive Position Change After Dimethicone Premedication Improves Gastric Cleanliness for Magnetically Controlled Capsule Endoscopy: a Single-blind, Randomized Controlled Trial
Brief Title: Repetitive Position Change Improves Gastric Cleanliness for MCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, M.D., Associate Professor, Associate Chief Physician, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MCE-RPC
Record Dates: First submitted 2018-04-17; First posted 2018-05-03 (Actual); Results first posted 2019-07-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Stomach Diseases
Keywords: Position change; Gastric cleanliness; Magnetically controlled capsule endoscopy
MeSH Terms: conditions — Stomach Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional group (No Intervention): Right after ingesting 5 g dimethicone mixed with 100 ml water, subjects in the conventional group will receive no intervention. Thirty and 40 min after dimethicone administration, subjects will additionally take 200 ml and 800 ml water, respectively, and undergo MCE examination.
- Position change group (Experimental): Right after ingesting 5 g dimethicone mixed with 100 ml water, subjects in the position change group will be instructed to repeatedly change the body position according to a pre-specified protocol for a period of 15 min: in the order of supine to the left lateral position to prone, left lateral, supine, right lateral, and repeat last four positions twice, each for 1 min; finally supine for 1 min. Thirty and 40 min after dimethicone administration, subjects in both groups will additionally take 200 ml and 800 ml water, respectively before undergoing MCE examination.
  Interventions: Behavioral: Position change group

INTERVENTIONS:
Behavioral: Position change group — Right after ingesting 5 g dimethicone mixed with 100 ml water, subjects in the position change group will be instructed to repeatedly change the body position according to a pre-specified protocol for a period of 15 min: in the order of supine to the left lateral position to prone, left lateral, supine, right lateral, and repeat last four positions twice, each for 1 min; finally supine for 1 min. Thirty and 40 min after dimethicone administration, subjects in both groups will additionally take 200 ml and 800 ml water, respectively before undergoing MCE examination.
  Arms: Position change group

SUMMARY:
By comparing dimethicone administration with/without subsequent repetitive position change before magnetically controlled capsule endoscopy (MCE) examination, the investigators aim to determine the efficacy of repetitive position change in improving gastric cleanliness for MCE examination.

DETAILED DESCRIPTION:
This is a single-blind, randomized controlled trial. Subjects receiving magnetically controlled capsule endoscopy at the institution will be randomly allocated into positional change group and conventional group before the procedure. Right after ingesting 5 g dimethicone mixed with 100 ml water, subjects in the position change group will be instructed to repeatedly change the body position according to a pre-specified protocol for a period of 15 min: in the order of supine to the left lateral position to prone, left lateral, supine, right lateral, and repeat last four positions twice, each for 1 min; finally supine for 1 min. Thirty and 40 min after dimethicone administration, subjects in both groups will additionally take 200 ml and 800 ml water, respectively, and undergo MCE examination. Gastric cleanliness will be rated by two physicians independently.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged more than 18 years, who were scheduled to undergo a magnetically controlled capsule endoscopy, were eligible for this study.

Exclusion Criteria:

* Dysphagia or symptoms of gastric outlet obstruction, suspected or known intestinal stenosis, overt gastrointestinal bleeding, history of upper gastrointestinal surgery or abdominal surgery altering gastrointestinal anatomy, or postabdominal radiation;
* Congestive heart failure, renal insufficiency, under therapeutic anticoagulation, in poor general condition (American Society of Anesthesiologists class III/IV), claustrophobia, metallic parts, a pacemaker or other implanted electromedical devices, artificial heart valves;
* Pregnancy or suspected pregnancy;
* Exclusion criteria for standard magnetic resonance imaging (MRI) examination such as the presence of surgical metallic devices, even though its low magnetic field would technically not interfere with such devices;
* Currently participating in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, Study Chair — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang YC, Pan J, Jiang X, Su XJ, Zhou W, Zou WB, Qian YY, Chen YZ, Liu X, Yu J, Yan XN, Zhao AJ, Li ZS, Liao Z. Repetitive Position Change Improves Gastric Cleanliness for Magnetically Controlled Capsule Gastroscopy. Dig Dis Sci. 2019 May;64(5):1297-1304. doi: 10.1007/s10620-018-5415-7. Epub 2018 Dec 17. PMID 30560329

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients with the following were excluded: (1) dysphagia or symptoms of gastric outlet obstruction; (2) poor general condition; (3) a pacemaker or other implanted electromedical devices, or artiﬁcial heart valves; (4) pregnancy or suspected pregnancy; (5) exclusion criteria for standard magnetic resonance imaging examination
Groups:
- Position Change Group: Right after ingesting 5 g dimethicone mixed with 100 ml water, subjects in the position change group were instructed by the study nurses to repeatedly change the body position according to a pre-specified protocol for a period of 15 min: in the order of supine position, left lateral position, three cycles of prone, left lateral, supine, and right lateral positions, and finally supine position, with a duration of 1 min for each position. Thirty and 40 min after dimethicone administration, subjects will additionally take 200 ml and 800 ml water, respectively before undergoing MCE examination.
Period: Overall Study
Arm/Group | Conventional Group | Position Change Group
Started | 40 | 43
Completed | 40 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects who met the inclusion criteria will be randomly allocated into position change or conventional groups. An independent research assistant generated the computerized random number sequence.
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Group | Position Change Group | Total
Number analyzed (Participants) | 40 | 43 | 83
Age, Continuous [Mean (Full Range); unit: years] | 45.3 [20 to 69] | 49.6 [22 to 80] | 47.5 [20 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 20 | 30
  Male | 30 | 23 | 53
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 40 | 43 | 93
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.6 (3.7) | 22.9 (3.1) | 23.9 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Image Cleanliness of Gastric Cavity
Description: The image cleanliness of gastric cavity of six primary anatomical landmarks of stomach (cardia, fundus, body, angulus, antrum, and pylorus) were recorded for evaluation. A 4-point grading scale was introduced to define the cleanliness as excellent (no adherent mucus and foam: score 4), good (mild mucus and foam but does not obscure vision: score 3), fair (considerable amount of mucus or foam present precluding a completely reliable examination: score 2) and poor (large amount of mucus or foam residue needing water to clear it: score 1)
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Conventional Group | Position Change Group
Number analyzed (Participants) | 40 | 43
units on a scale
  cardia | 3.0 (0.6) | 3.5 (0.5)
  fundus | 2.2 (0.7) | 3.0 (0.6)
  body | 2.7 (0.7) | 3.1 (0.4)
  angulus | 3.1 (0.7) | 3.7 (0.5)
  antrum | 3.7 (0.5) | 4.0 (0.0)
  pylorus | 3.9 (0.3) | 4.0 (0.0)

2. Secondary Outcome: The Type of Positive Findings Detected by Magnetically Controlled Capsule Gastroscopy
Description: Positive findings defined as any pathology detected by Magnetically controlled capsule gastroscopy (MCCG), including polyps, ulcer, gastric fundus varices, submucosal tumor, and carditis.
Time Frame: 30 minutes
Measure: Number; unit: findings
Arm/Group | Conventional Group | Position Change Group
Number analyzed (Participants) | 40 | 43
findings | 11 | 12

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Safety of MCCG, or adverse events, defined as symptoms or signs such as abdominal distention, nausea, or vomiting, were monitored closely during the MCCG procedure. Capsule retention (i.e., a capsule endoscope remaining in the gastrointestinal tract for more than two weeks or a capsule endoscope that requires directed intervention or therapy to aid its expulsion) was monitored and followed up for up to two weeks.
Time Frame: 2 weeks
Measure: Number; unit: participants
Arm/Group | Conventional Group | Position Change Group
Number analyzed (Participants) | 40 | 43
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Safety of MCCG, or adverse events, defined as symptoms or signs such as abdominal distention, nausea, or vomiting, were monitored closely during the MCCG procedure. Capsule retention (i.e., a capsule endoscope remaining in the gastrointestinal tract for more than two weeks or a capsule endoscope that requires directed intervention or therapy to aid its expulsion) was monitored and followed up for up to two weeks.
Groups:
- Conventional Group: Right after ingesting 5 g dimethicone mixed with 100 ml water, subjects in the conventional group will receive no intervention. Thirty and 40 min after dimethicone administration, subjects will additionally take 200 ml and 800 ml water, respectively, and undergo MCCG examination.
- Position Change Group: Right after ingesting 5 g dimethicone mixed with 100 ml water, subjects in the position change group will be instructed to repeatedly change the body position according to a pre-specified protocol for a period of 15 min: in the order of supine to the left lateral position to prone, left lateral, supine, right lateral, and repeat last four positions twice, each for 1 min; finally supine for 1 min. Thirty and 40 min after dimethicone administration, subjects in both groups will additionally take 200 ml and 800 ml water, respectively before undergoing MCCG examination.
Arm/Group | Conventional Group | Position Change Group
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/43
Other Adverse Events (participants affected / at risk) | 0/40 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT03514966/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-01): https://cdn.clinicaltrials.gov/large-docs/66/NCT03514966/SAP_001.pdf